CLINICAL TRIAL: NCT01628081
Title: A Randomized, Double-Blind, , Placebo Controlled, 18 Week Study To Evaluate the Efficacy of Adjuvant 9-cis-β-Carotene Rich Powder of the Alga Dunaliella Bardawil in Subjects With Plaque Type Psoriasis.
Brief Title: The Effect of Alga Dunaliella Bardawil on Psoriasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHEBA-12-9174-SG-CTIL
Record Dates: First submitted 2012-06-14; First posted 2012-06-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Psoriasis
Keywords: psoriasis; Alga Dunaliella Bardawil
MeSH Terms: conditions — Psoriasis | interventions — Cbr protein, Dunaliella

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alga Dunaliella bardawil (Experimental): After screen phase of maximum two weeks the subjects will be randomized to one of two treatments groups (1:1): Dunaliella or placebo.
  Interventions: Dietary Supplement: Dunaliella Bardawil
- Placebo (Placebo Comparator): Dosage Regimen and Treatment Groups
  * Daily oral administration of:
  * Dunaliella, 6 capsules/day (3 capsules in the morning, 3 in the evening).
  * Placebo, 6 capsules/day (3 capsules in the morning, 3 in the evening).
  Interventions: Dietary Supplement: Alga Dunaliella Bardawil placebo

INTERVENTIONS:
Dietary Supplement: Alga Dunaliella Bardawil placebo — Dosage Regimen and Treatment Groups
  * Daily oral administration of:
  * Dunaliella, 6 capsules/day (3 capsules in the morning, 3 in the evening).
  * Placebo, 6 capsules/day (3 capsules in the morning, 3 in the evening).
  Arms: Placebo
Dietary Supplement: Dunaliella Bardawil — Dosage Regimen and Treatment Groups
  * Daily oral administration of:
  * Dunaliella, 6 capsules/day (3 capsules in the morning, 3 in the evening).
  * Placebo, 6 capsules/day (3 capsules in the morning, 3 in the evening).
  Arms: Alga Dunaliella bardawil

SUMMARY:
This is a double blind, parallel group, randomized study with 12 weeks of daily oral administration of Dunaliella or placebo in psoriasis patients.

DETAILED DESCRIPTION:
Subjects will be screened for eligibility at the baseline visit for blood tests.

After screen phase of maximum two weeks the subjects will be randomized to one of two treatments groups (1:1): Dunaliella or placebo.

Each subject will have a final evaluation 4 weeks after the end of study drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, ≥ 18 to ≤ 75 years of age, who have a diagnosis of plaque or guttate psoriasis;
* Psoriasis covering ≤ 20% of body surface area (BSA)
* Have at least 2 psoriatic plaques measuring 3 cm or more.
* For a female subject; either:
* subject is non-childbearing potential, defined as: menopause with amenorrhea > 2 years, hysterectomy, or bilateral oophorectomy or
* agrees to continue to use adequate contraception (i.e., hormonal [oral, depot, patch], IUD, barrier and spermicide) throughout the study and for at least one month following termination and have a negative urinary pregnancy test at screening and before the first dose of study drug;
* In the opinion of the Investigator, the subject will be compliant and have a high probability of completing the study and all required procedures.

Exclusion Criteria:

* The subject presents with the predominant type of psoriasis as erythrodermic, inverse, pustular or palmo-plantar or an unstable form of psoriasis;
* Received any investigational drug within 30 days of randomization.
* The subject has not used the following psoriasis treatment for the elaborated periods, prior to the date of screening visit:

Topical psoriasis treatment, excluding emollients 2-week period Any systemic psoriasis treatment including biologic treatments 4-week or 5-half life time periods (whichever is longer) Phototherapy or Climatotherapy 4-week period

* The subject has a known allergy or sensitivity to the study treatment(s) or to any of the percipient contained in the study drug formulation
* Any other acute or chronic medical condition that, in the opinion of the Investigator, increases the risk to the subject or the likelihood that the subject will be unable to complete the study;
* Subjects with any laboratory test at screening considered significantly abnormal.

The following will be considered significantly abnormal:

Alanine transaminase (ALT), aspartate transaminase (AST) > 3 upper limit normal. CPK > 3 upper limit normal. Triglycerides > 350mg/dl.

cytopenia (to include any of the following: WBC < 35000/μL; Hgb < 10 g/dL; platelets <120,000/μL; neutrophils absolute < 1500/μL lymphocytes absolute < 800/μL) or

* Known serologic positively for human immunodeficiency virus or hepatitis B or hepatitis C virus.
* History of substance abuse, including alcohol abuse, within the past year.
* History or current clinically significant major psychiatric disorder (e.g., major depressive disorder, psychosis, schizophrenia) according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM IV TR) [Exception; subjects with depression that has been adequately controlled for at least 6 months may enroll in the study];
* Female subject with a positive pregnancy test or nursing, or planning a pregnancy during the course of the study;
* Unwilling or unable to comply with study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline (predose day 1) to 18-week period Target Lesion Severity score (TLS) of lesions | Subjects will have study visits at screening- visit 1, randomization - visit 2, after 6 weeks treatment - visit 3, 12 weeks treatment -end of treatment - visit 4 and week 16 - follow up visit 5.
  Target lesions will be evaluated for 3 components: erythema, induration, and scaling. Each component will be given a score using the following scale: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. The Target Lesion Severity (TLS) score is calculated as a sum of the 3 components.

CONTACTS AND LOCATIONS:
Overall Officials: Shoshana Greenberg, MD, Principal Investigator — Sheba Medical Center
Locations (2):
- Israel (2):
  - The Bert W. Strassburger Lipid Center,Sheba Medical Center, Tel Litwinsky
  - The Bert W. Strassburger Lipid Center, Tel Litwinsky